CLINICAL TRIAL: NCT03779451
Title: Vaginal Progesterone Versus 17-Alpha-Hydroxyprogesterone Caproate for Prevention of Emergent Cesarean Delivery in Asymptomatic Pregnant Women With Placenta Previa: A Randomized Controlled Study
Brief Title: Vaginal Progesterone Versus 17-Alpha-Hydroxyprogesterone Caproate in Placenta Previa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: aswu/191/18
Record Dates: First submitted 2018-12-15; First posted 2018-12-19 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Placenta Previa
Keywords: cesarean section; placenta previa; antepartum hemorrhage; vaginal progesterone; 17-Alpha-Hydroxyprogesterone Caproate
MeSH Terms: conditions — Placenta Previa | interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: A randomized controlled study
Masking Description: An open-label randomized controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 17-OHPC (Active Comparator): patients received weekly 250 mg 17 alpha-hydroxyprogesterone-caproate (cidolut depot) intramuscular injections started at 26-28 week and up to 37-weeks' gestation or delivery
  Interventions: Drug: 17-OHPC
- vaginal progesterone (Active Comparator): vaginal progesterone suppositories (Cyclogest vaginal suppository) in a dose of 400 mg daily at bedtime starting at 26-28 weeks of gestation till 37 weeks of gestation or delivery
  Interventions: Drug: vaginal progesterone
- control group (No Intervention): Women with gestational age from 26-28 weeks diagnosed with placenta previa who will not receive vaginal progesterone.

INTERVENTIONS:
Drug: 17-OHPC — received weekly 250 mg 17 alpha-hydroxyprogesterone-caproate (cidolut depot) intramuscular injections started at 26-28 week and up to 37-weeks' gestation or delivery.
  Other Names: Active Comparator; cidolut depot
  Arms: 17-OHPC
Drug: vaginal progesterone — vaginal progesterone suppositories (Cyclogest vaginal suppository) in a dose of 400 mg daily starting at 26-28 weeks of gestation till 37 weeks of gestation or delivery
  Other Names: Active Comparator; Cyclogest
  Arms: vaginal progesterone

SUMMARY:
Purpose to evaluate the effects of Vaginal Progesterone versus 17-Alpha-Hydroxyprogesterone Caproate for prevention of Emergent Cesarean Delivery in Asymptomatic Pregnant Women with Placenta Previa

DETAILED DESCRIPTION:
The study will be a randomized open-label clinical trial conducted at a tertiary university hospital outpatient clinic and some private settings at Aswan governorate, Egypt, between January 2019 and March 2022. The authors will include women who asymptomatic pregnant women with a diagnosed placenta previa at 26-28 weeks gestation. They will be randomized into three groups: group I (vaginal progesterone suppositories ), group II (received an intramuscular dose of 250 mg 17-alpha-Hydroxyprogesterone caproate(17-OHPC) once a week) and group III(control group). In each group, Follow-up visits were performed every week then admission was done at 36 weeks at our university hospital. Scheduled caesarian section was done at completed 37 weeks unless otherwise required.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 26-28 weeks of gestation.
* Definite and reliable diagnosis of placenta previa (defined as the presence of a placenta within 2 cm of the internal os), using a transvaginal ultrasound scan

Exclusion Criteria:

* Multiple pregnancies.
* Women at high risk of preterm labor e.g. history of spontaneous preterm labor or preterm prelabour rupture of the membranes (PPROM).
* Severe antepartum hemorrhage and/or hemodynamic instability that necessitates urgent -intervention and delivery.
* Women who have been maintained on progestin therapy since early pregnancy for whatever reason.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women with placenta previa
Enrollment: 400 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
number of patient delivered before 37 weeks | 2 month
  calculation the number of patients delivered before 37 weeks

SECONDARY OUTCOMES:
number of episodes of antepartum hemorrhage | 2 month
  calculating the mean number of episodes of antepartum hemorrhage
Hospital admission for significant antepartum hemorrhage | 2 month
  Number of patients requiring hospital admission for significant antepartum hemorrhage
Neonatal Birth weight | one hours post operative
  measure Neonatal Birth weight in kilograms

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided